CLINICAL TRIAL: NCT05138900
Title: A Pilot Study of Single Fraction Stereotactic Body Radiation Therapy (SBRT) in Central Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 1307721
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiation Therapy (SBRT) (Experimental): A single fraction of targeted SBRT
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — SBRT for central non small cell lung cancer
  Other Names: Stereotactic Body Radiation Therapy

SUMMARY:
The purpose of this study is to determine if a single treatment of targeted radiation (called SBRT or Stereotactic Body Radiation Therapy) can be as safe and effective as multiple doses of radiation in patients with central non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Have an ECOG Performance Status of ≤ 2. Refer to Appendix A.
* Have histologically proven diagnosis of non-small cell lung cancer (NSCLC).
* Stage cT1-3N0M0 with tumor size < 6 cm.
* Prior systemic therapy allowed but no systemic therapy 4-6 weeks prior to stereotactic body radiation therapy SBRT (see exclusion criteria), during SBRT, or 2 weeks after SBRT.
* Tumors located within 2 cm in all directions of any mediastinal critical structures, including the bronchial tree, esophagus, heart, brachial plexus, major vessels, spinal cord, phrenic nerve, and recurrent laryngeal nerve, as defined by the International Association for the Study of Lung Cancer (IASLC) (27).
* Participant is considered to be either medically or surgically inoperable by physicians, or participant declines surgery.
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry.

Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Contraindication to stereotactic body radiation therapy (SBRT) (including the inability to cooperate with any aspect of SBRT such as the inability to lie still and breathe reproducibly)
* Prior radiation to the volume of lung or mediastinum currently involved by tumor
* Plan for the patient to receive other concomitant antineoplastic therapy (including standard fractionated radiation, chemotherapy, biological therapy, vaccine therapy, and surgery) while on this protocol, except at disease progression
* Received an investigational agent within 30 days prior to enrollment
* Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female participants.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive SBRT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2028-03-09 (Estimated); Study Completion 2028-03-09 (Estimated)

PRIMARY OUTCOMES:
Rate of grade 3-5 adverse events | Up to 5 years
  Rates of treatment related grade 3-5 adverse events. Assessed using CTCAE v.5

SECONDARY OUTCOMES:
Progression-free Survival | Up to 5 years
  Progression free is defined as time from initiation of SBRT to disease progression or death from any cause. Estimated by the Kaplan-Meier method.
Overall Survival | UP to 5 years
  Overall Survival is defined as time from initiation of SBRT to patient death from any cause. Estimated by the Kaplan-Meier method.
Quality of life scores | Up to 5 years
  Comparison of QoL scores between time points will be made using the Wilcoxon signed rank test
Local Control Rate | Up to 5 years
  Local control is defined as absence of local failure among patients evaluable for efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided